CLINICAL TRIAL: NCT04603833
Title: A Phase II Clinical Study of SHR3680 Combined With Docetaxel in the Treatment of Metastatic Castration-resistant Prostate Cancer Previously Treated With Abiraterone
Brief Title: A Study of SHR3680 in Combination With Docetaxel in the Treatment of mCRPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR3680-II-203
Record Dates: First submitted 2020-10-22; First posted 2020-10-27 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-10

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR3680+Docetaxel (Experimental)
  Interventions: Drug: SHR3680+Docetaxel
- SHR3680 (Active Comparator)
  Interventions: Drug: SHR3680
- Docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: SHR3680+Docetaxel — Participants will receive SHR3680 combined with Docetaxel
  Arms: SHR3680+Docetaxel
Drug: SHR3680 — Participants will receive SHR3680
  Arms: SHR3680
Drug: Docetaxel — Participants will receive Docetaxel
  Arms: Docetaxel

SUMMARY:
The aim of this trial is to evaluate SHR3680 combined with Docetaxel to improve Metastatic Castration Resistant Prostate Cancer Patients whether the patient's Time to prostate specific antigen (PSA) progression is superior to SHR3680 or Docetaxel single drug.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed prostate cancer; Unconfirmed neuroendocrine carcinoma or small cell carcinoma;
2. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1;
3. Radiographic evidence of metastasis（CT/MRI/ECT);
4. Sustained therapy of luteinizing hormone-releasing hormone analogue(LHRHA)or received bilateral orchiectomy; patients who did not receive bilateral orchiectomy are willing to receive sustained therapy of LHRHA;
5. Evidence of prostate cancer progression under the sustained therapy of LHRHA or bilateral orchiectomy;
6. Adequate hepatic, renal, heart, and hematological functions;
7. Patients have given voluntary written informed consent before performance of any study-related procedure not part of normal medical care,with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care；
8. Expected to survive for at least 3 months；
9. Patient has been treated with Abiraterone and treatment failed；Treatment failure is defined as the progression of disease during treatment；

Exclusion Criteria:

1. Have received any anti-tumor therapy in the past 4 weeks,including radiotherapy, chemotherapy, operation, targeted therapy, immuntherapy, and endocrinotherapy;
2. As a subject to participate in other drug clinical trials, the last test drug was administered within 4 weeks from the first dose of the study drug;
3. Plan to receive any other anti-tumor treatment during this trial;
4. Subjects have contraindications to prednisone, such as active infections or other conditions;
5. Subjects present any chronic condition requiring treatment with corticosteroids at doses greater than prednisone 5 mg, BID;
6. The investigators judged severe bone damage caused by tumor bone metastasis, including severely controlled bone pain, pathological fractures and spinal cord compressions that occurred in the last 6 months or are expected to occur in the near future;
7. Uncontrolled high blood pressure (systolic blood pressure 160 mmHg or diastolic blood pressure 95 mmHg). If blood pressure can be effectively controlled by antihypertensive therapy, subjects with a history of hypertension are allowed to participate in the study;
8. Study of active heart disease within 6 months prior to the first dose, including: severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, left ventricular ejection fraction <50%, and room for medication Arrhythmia;
9. Imaging diagnosis of brain tumor lesions;
10. history of pituitary or adrenal dysfunction;
11. Study of other malignant tumors within 5 years prior to the first dose (in situ cancer with complete remission and excluding malignant tumors with slow progress);
12. Patients with active HBV or HCV infection (HBV virus copy number #104 copies/mL, HCV virus copy number #103 copies/mL), or active syphilis infection;
13. History of immunodeficiency (including HIV positive, other acquired, congenital immunodeficiency disease) or organ transplant history;
14. Habitual constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease; abdominal fistula, gastrointestinal perforation or abdominal abscess within 6 months before the first dose;
15. Patients who are unwilling to take effective contraceptive measures during the entire study period and within 3 months after the last dose

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to prostate specific antigen (PSA) progression | [Time Frame: Approximately 24 months]
  Time from randomisation to the first time of PSA progression according to the criterion of PCGW3
Adverse Event(AE) | [Time Frame: Approximately 24 months]
  The type, frequency, severity, timing, seriousness, and relationship to study therapy

SECONDARY OUTCOMES:
Radiographic Progression Free Survival(rPFS) | [Time Frame: Approximately 24 months]
  Time from randomisation to radiologically confirmed progressive disease or death due to any cause
Objective response rate (ORR) | [Time Frame: Approximately 24 months]
  The percentage of patients with measureable disease at baseline who achieved a complete or partial response in their soft tissue disease using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria
PSA response rate | [Time Frame: Approximately 3 months]
  After the continuous therapy from randomisation to the end of the 12 weeks, the percentage of patients whose levels of PSA decreased by more than 50% compared with baseline
Overall Survival(OS) | [Time Frame: Approximately 24 months]
  Time from randomisation to death due to any cause
Area Under the Curve (AUC) | [Time Frame: Approximately 2 months]
  The single dose and multiple dose PK will be calculated as data permits including AUC
Maximum Observed Plasma Concentration (Cmax) | [Time Frame: Approximately 2 months]
  The single-dose and multiple dose PK will be calculated as data permits including Cmax
Minimum Observed Plasma Concentration (Cmin) | [Time Frame: Approximately 2 months]
  The single-dose and multiple dose PK will be calculated as data permits including Cmin

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No